CLINICAL TRIAL: NCT03279679
Title: A Randomized Comparison of Minimum Effective Volume With 0.5% Ropivacaine Between Costoclavicular and Paracoracoid Ultrasound-guided Infraclavicular Block for Forearm Surgery
Brief Title: Comparison Between Costoclavicular and Paracoracoid Ultrasound-guided Infraclavicular Block for Forearm Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, PhD, MD Vice-Director of Anestheiology Department, Tongji hospital, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB20170702
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Brachial Plexus Block
Keywords: costoclavicular; paracoracoid; brachial plexus
MeSH Terms: interventions — Ultrasonography; Ropivacaine

STUDY DESIGN:
Intervention Model Description: costoclavicular group and paracoracoid group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- costoclavicular group (Experimental): patients in this group are assigned to receive ultrasound-guided costoclavicular infraclavicular block with 0.5% ropivacaine for upper limb surgery at elbow joint and below
  Interventions: Procedure: costoclavicular infraclavicular block; Device: Ultrasound; Drug: Ropivacaine
- paracoracoid group (Other): patients in this group are assigned to receive ultrasound-guided paracoracoid infraclavicular block with 0.5% ropivacaine for upper limb surgery at elbow joint and below
  Interventions: Procedure: paracoracoid infraclavicular block; Device: Ultrasound; Drug: Ropivacaine

INTERVENTIONS:
Procedure: costoclavicular infraclavicular block — Infraclavicular brachial plexus block will be performed through new costoclavicular space approach under realtime ultrasound guidance with 0.5% ropivacaine
  Arms: costoclavicular group
Procedure: paracoracoid infraclavicular block — Infraclavicular brachial plexus block will be performed through traditional paracoracoid approach under realtime ultrasound guidance with 0.5% ropivacaine
  Arms: paracoracoid group
Device: Ultrasound — All the nerve blocks will be performed under realtime ultrasound guidance
Drug: Ropivacaine — 0.5% ropivacaine will be used for the brachial plexus block in both groups.

SUMMARY:
The costoclavicular space block technique is a new developed approach of ultrasound-guided infraclavicular brachial plexus block(USG-ICB) in last two years and has not been studied much yet. The paracoracoid approach serves as a standard and traditional method for USG-ICB in clinical practice, easy to learn and perform. The investigators set this parallel controlled dose-finding trial to work out the MEV with 0.5% ropivacaine of both two approaches above for forearm surgery and compare the performance time between them, providing reasonable evidence for clinical choice.

DETAILED DESCRIPTION:
The costoclavicular space block technique is a new developed approach of ultrasound-guided infraclavicular brachial plexus block(USG-ICB) in last two years and has not been studied much yet. USG-ICB represents an attractive option for upper-limb surgery at or below the elbow joint with similar success rate and fewer adverse effects compared with ultrasound-guided supraclavicular block. The paracoracoid approach serves as a standard and traditional method for USG-ICB in clinical practice, easy to learn and perform. However, the minimum effective volume(MEV)of this approach has been studied by different investigators with different regional anesthetics or its mixture, and specially, the 95% MEV result of this approach is more than 30ml in all related researches which is still a large volume. According to the investigators' experience in using the costoclavicular space technique for forearm surgery, it usually can get a comparable sensation and motor block effect by no more than 25ml. Recently, there was a clinical randomized control study which compared the costoclavicular and paracoracoid USG-ICB for upper limb surgery using a 35ml-mixture of 1% lidocaine-0.25% bupivacaine with epinephrine 5 ug/ml and came to the conclusions: two groups resulted in similar onset times and no intergroup difference were found in terms of performance time and success rate. However, 35ml is a much larger regional anesthetic volume than what we used in routine brachial plexus block. So, we set this parallel controlled dose-finding trial to work out the MEV with 0.5% ropivacaine of both approaches above for forearm surgery and compare the performance time between them, providing reasonable evidence for clinical choice. Patients enrolled in this study will be assigned to costoclavicular group and paracoracoid group and in each group, the volume of local anesthetic applied to patients start with 30ml, and then decreased by 2.5ml for next patient when the previous block is successful, otherwise increased by 2.5ml when failed,which is also called a staircase up-and-down method usually applied in dose-finding research of nerve block. After certain reflections of the local anesthetic volume sequential line graph, the minimum effective volume could be calculated.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1 to 3
* BMI 20-35
* Scheduled for surgery at elbow joint or below

Exclusion Criteria:

* Inability to consent to the study
* Preexisting neuropathy,coagulopathy,COPD
* Hepatic or renal failure
* Allergy to local anesthetics
* Pregnancy
* Prior surgery in infraclavicular region

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
MEV | The anesthesia effect of the block with a specified volume fo local anesthetic will be assessed at 30 min after the nerve block finished, the MEV will be calculated after all.
  minimum effective volume regional anesthetic need for a successful infraclavicular block

SECONDARY OUTCOMES:
performance time | from the time point when ultrasound probe touches with patients' skin to the end when local anesthetic is injected through the needle, which is usually up to ten minutes
  time needed for the block performance

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, MD, Study Director — Department of anesthesiology, Tongji hospital, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrecht E, Mermoud J, Fournier N, Kern C, Kirkham KR. A systematic review of ultrasound-guided methods for brachial plexus blockade. Anaesthesia. 2016 Feb;71(2):213-27. doi: 10.1111/anae.13347. Epub 2015 Dec 16. PMID 26670119
- [Background] Park SK, Lee SY, Kim WH, Park HS, Lim YJ, Bahk JH. Comparison of Supraclavicular and Infraclavicular Brachial Plexus Block: A Systemic Review of Randomized Controlled Trials. Anesth Analg. 2017 Feb;124(2):636-644. doi: 10.1213/ANE.0000000000001713. PMID 27828793
- [Background] Sauter AR, Smith HJ, Stubhaug A, Dodgson MS, Klaastad O. Use of magnetic resonance imaging to define the anatomical location closest to all three cords of the infraclavicular brachial plexus. Anesth Analg. 2006 Dec;103(6):1574-6. doi: 10.1213/01.ane.0000242529.96675.fd. PMID 17122242
- [Background] Tran DQ, Dugani S, Dyachenko A, Correa JA, Finlayson RJ. Minimum effective volume of lidocaine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):190-4. doi: 10.1097/AAP.0b013e31820d4266. PMID 21270721
- [Background] Tran DQ, Bertini P, Zaouter C, Munoz L, Finlayson RJ. A prospective, randomized comparison between single- and double-injection ultrasound-guided infraclavicular brachial plexus block. Reg Anesth Pain Med. 2010 Jan-Feb;35(1):16-21. doi: 10.1097/AAP.0b013e3181c7717c. PMID 20048654
- [Background] Flohr-Madsen S, Ytrebo LM, Kregnes S, Wilsgaard T, Klaastad O. Minimum effective volume of ropivacaine 7.5 mg/ml for an ultrasound-guided infraclavicular brachial plexus block. Acta Anaesthesiol Scand. 2013 Apr;57(4):495-501. doi: 10.1111/aas.12078. Epub 2013 Feb 18. PMID 23418881
- [Background] Sala-Blanch X, Reina MA, Pangthipampai P, Karmakar MK. Anatomic Basis for Brachial Plexus Block at the Costoclavicular Space: A Cadaver Anatomic Study. Reg Anesth Pain Med. 2016 May-Jun;41(3):387-91. doi: 10.1097/AAP.0000000000000393. PMID 27035461
- [Background] Leurcharusmee P, Elgueta MF, Tiyaprasertkul W, Sotthisopha T, Samerchua A, Gordon A, Aliste J, Finlayson RJ, Tran DQH. A randomized comparison between costoclavicular and paracoracoid ultrasound-guided infraclavicular block for upper limb surgery. Can J Anaesth. 2017 Jun;64(6):617-625. doi: 10.1007/s12630-017-0842-z. Epub 2017 Feb 15. PMID 28205117
- [Background] Petrar SD, Seltenrich ME, Head SJ, Schwarz SK. Hemidiaphragmatic paralysis following ultrasound-guided supraclavicular versus infraclavicular brachial plexus blockade: a randomized clinical trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):133-8. doi: 10.1097/AAP.0000000000000215. PMID 25650633